CLINICAL TRIAL: NCT06687694
Title: Immune Mechanisms of Antipsychotic Treatment Response
Acronym: IMAT
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other); University of Oxford (Other); McPin Foundation (Other); Francis Crick Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 331728
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Psychosis
Keywords: Psychosis; Antipsychotic; Neuroimmunology; Inflammation; Autoantibody; Schizophrenia; Schizotypal disorder; Persistent delusional disorders; Acute and transient psychotic disorders; Induced delusional disorder; Schizoaffective disorders; Other nonorganic psychotic disorders; Unspecified nonorganic psychosis; Manic episode; Bipolar affective disorder; Depressive episode; Recurrent depressive disorder; Persistent mood [affective] disorders; Other mood [affective] disorders; Unspecified mood [affective] disorder
MeSH Terms: conditions — Psychotic Disorders; Inflammation; Schizophrenia; Schizotypal Personality Disorder; Shared Paranoid Disorder; Mental Disorders; Mania; Bipolar Disorder; Depressive Disorder; Mood Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and cerebrospinal fluid.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Participants with psychosis symptoms
- Control Participants

SUMMARY:
The aim of this study is to investigate the role of the immune system in psychotic symptoms and their response to treatment. The investigators will collect blood and cerebrospinal fluid samples from participants with psychosis symptoms who are about to start or change to a new regular antipsychotic treatment as well as a control group for comparison.

Participants will be assessed at two main timepoints, at visit 1 (Week 0) and at visit 2 (4 +/-2 weeks). For participants with psychosis symptoms visit 1 will take place at the start or change of antipsychotic medication. The studies goal is to identify biomarkers that can aid in diagnosis, prognosis, treatment selection, and tracking treatment response.

The investigators aim to recruit participants from the following groups:

1. Individuals with psychosis symptoms presenting to acute or outpatient services who are due to be started on or change to a new regular antipsychotic medication.
2. Age- and sex-matched control participants without neuropsychiatric disease.

Findings could potentially impact the treatment of psychotic illnesses by offering mechanistic insights into targeted immune-based interventions for these disorders through high-resolution immunophenotyping techniques alongside targeted immunological assays. Ultimately, the research aims to contribute valuable resources for future studies exploring the connection between immune processes and neuropsychiatric conditions.

ELIGIBILITY:
Inclusion Criteria

Participants with psychosis symptoms:

* Age 18-65
* Currently experiencing psychosis symptoms warranting treatment by secondary care mental health services, as confirmed by a psychiatrist involved in their treatment.
* Psychosis symptoms likely to be attributable to a disorder represented by ICD codes F20-F39, in the opinion of the treating clinical team.
* Due to start or change to a new regular antipsychotic medication. (Participants who are initiating antipsychotic treatment for the first time, transitioning to a different antipsychotic medication, or resuming a formerly prescribed antipsychotic medication that was discontinued for a minimum of two weeks may be recruited.)

Control Participants

* Age 18-65
* No active autoimmune disorder.
* No history of psychosis symptoms.

Exclusion Criteria

Participants with psychosis symptoms:

* Unacceptable risk of harm to participant or study staff due to risk of behavioural disturbance.
* Currently taking or having taken in the last four weeks any medication known to grossly affect the production or function of immune cells (e.g. corticosteroids, methotrexate, cyclophosphamide, mycophenolate mofetil, rituximab or other monoclonal antibody therapies).
* Inability to have blood tests.

Control participants:

* Unacceptable risk of harm to participant or study staff due to risk of behavioural disturbance.
* Currently taking or having taken in the last four weeks any medication known to grossly affect the production or function of immune cells (e.g. corticosteroids, methotrexate, cyclophosphamide, mycophenolate mofetil, rituximab or other monoclonal antibody therapies).
* Inability to have blood tests.

Optional lumbar puncture only:

* Significant lower spinal deformity (such as spina bifida), injury (such as stenosis) or previous lower spinal surgery.
* Antiplatelet or anticoagulant therapy within the 14 days prior to Lumbar Puncture procedure.
* Known or suspected clotting disorder.
* Clinically significant abnormality in full blood count.
* Known or suspected raised intracranial pressure, assessed by study clinician.
* Known or suspected allergy to local anaesthetic agent or an ingredient of the anaesthetic solution.
* History of chronic or recurrent headaches, in the opinion of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with psychosis symptoms will be recruited from clinical services at participating sites. Control participants may be recruited via online and offline channels. This may include posting on social media platforms, sharing information with local research networks or databases and displaying adverts on notice boards in public places in collaborating universities and NHS facilities.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2031-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Peripheral Immune Phenotype | 4 +/-2 weeks
  Change in the flow cytometric peripheral immune phenotype following treatment with antipsychotic medication.

CONTACTS AND LOCATIONS:
Locations (1):
- South London and Maudsley NHS Foundation Trust, London, United Kingdom, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided